CLINICAL TRIAL: NCT00539071
Title: High Dose Risperidone Consta for Patients With Schizophrenia With Unsatisfactory Response to Standard Dose Risperidone or Long-Acting Injectable
Brief Title: High Dose Risperidone Consta for Patients With Schizophrenia With Poor Response to Risperidone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070580
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2025-08-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; long acting injectable; treatment resistant
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional dose (Active Comparator): All of those who are randomized to the conventional Consta dose will receive it in the form of Consta at a starting dose of 50 mg q 2 weeks (given as two injections - active 50 mg plus placebo injection).As advised by the package insert for Consta, oral risperidone will be given (3-4 mg qd x 3 days followed by 6mg qd up to Week 3 unless symptoms warrant a quicker titration) along with the injections.Any oral risperidone the patients receive will be discontinued after Week 4.At Week 6, psychopathology will be assessed with a PANSS. Dose will remain at 50 mg q 2 weeks for those in the conventional Consta dose group.
  Interventions: Drug: long-acting injectable risperidone; Drug: long acting injectable risperidone, Conventional Dose Group
- High Dose group (Active Comparator): Those who are randomized to high dose Consta will receive Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose after consent. As advised by the package insert for Consta, oral risperidone will be given (3-4 mg qd x 3 days followed by 6mg qd up to Week 4 unless symptoms warrant a quicker titration) along with the injections. Any oral risperidone the patients receive will be discontinued after Week 4.Psychopathology will be assessed with a PANSS at Week 6. If no improvement since baseline, dose will be increased to two 50 mg injections q 2 weeks for the remainder of the study.
  Interventions: Drug: long-acting injectable risperidone; Drug: long acting injectable risperidone, High Dose Group

INTERVENTIONS:
Drug: long-acting injectable risperidone — Subjects will be randomized to conventional dose Consta or high dose Consta. All of those who are randomized to the conventional Consta dose will receive it in the form of Consta at a starting dose of 50 mg q 2 weeks. Those who are randomized to high dose Consta will receive a Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose.Oral risperidone will be given up to Week 4 along with the injections for both groups to provide a transition phase.At Week 6, psychopathology will be assessed with a PANSS. If no improvement from baseline is shown, the randomized dose of Consta will be increased to 100 mg q 2 weeks (given as two 50 mg injections ) for those in the high dose Consta group. The dose for those randomized to the conventional dose group will remain the same (50 mg plus placebo).
Drug: long acting injectable risperidone, Conventional Dose Group — Study dose remains 50 mg for the length of the study.
  Other Names: Risperidone Consta/Conventional Dose
  Arms: Conventional dose
Drug: long acting injectable risperidone, High Dose Group — Beginning dose 75 mg. Can be increased to 100 mg at Week 6.
  Other Names: Risperidone Consta/High Dose
  Arms: High Dose group

SUMMARY:
The purpose of this study is to look at two doses of long-acting injectable risperidone (Risperdal Consta). The study will use a usual dose of Risperdal Consta (50 mg given every two weeks) or a higher dose (75 mg-100 mg given every two weeks) to see which one is better at improving symptoms of schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
This six month double-blind,randomized trial is designed to compare the efficacy of high dose long acting risperidone ( 75 mg-100 mg q2 weeks or its equivalent) with standard doses of long acting risperidone (≤50 mg/q 2weeks) for Total Psychopathology, positive, negative, and depressive symptoms, and cognition in patients who are considered to be poor responders by themselves, significant others, or clinicians. This will include two types of inadequately responding patients-those who are treatment resistant by research criteria (Kane et al., 1988) and those with inadequate response

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia or schizoaffective disorder
* Able to give written informed consent.
* Moderate psychosis persists although compliant with medication
* Patients must have an inadequate response to two antipsychotic medications (can be risperidone, oral or long acting - but not required), at doses that are within the upper end of the standard dosage range
* Patients must have a Clinical Global Impression - Severity (CGI-S) scale score at screening of at least moderate severity and a Personal and Social Performance Scale (PSP) score of 60 or below.
* At the time of screening, eligible patients will be receiving or have received treatment with risperidone oral or Consta, or a combination that does not exceed 50 mg q 2 weeks of Consta or oral risperidone 8 mg/day for at least 6 weeks within seven years of study entry without satisfactory response as documented in the medical record Risperidone
* Patients who have received Consta injectable medication within the specified dose range for no more than a month prior to the onset of the study will be eligible. Patients receiving mood stabilizers or antidepressants, or both, in addition to risperidone oral or Consta, will be eligible
* Patients may initially be inpatients or outpatients
* Females of childbearing potential will be admitted only if they are on stable birth control medication and understand that they should not get pregnant during the course of the study.
* All patients must have stable housing at the current time or plans for housing following hospital discharge, if an inpatient.
* Patients must be willing to receive injectable medication

Exclusion Criteria:

* Patients with a diagnosis other than schizophrenia or schizoaffective disorder.
* Patients previously treated with doses of these agents higher than those allowed for at least six months and who failed to have an adequate response will be excluded
* Patients currently taking clozapine or have failed an adequate trial of clozapine which lasted at least 3 months
* Pregnant females. Females who are currently breastfeeding will be excluded.
* Patients with a diagnosis of substance dependence at screening or up to one year prior to enrollment.
* Patient with worse than mild tardive dyskinesia or history of marked Extrapyramidal Symptoms (EPS) at screening
* Patients who have had neuroleptic malignant syndrome
* Patients with a history of galactorrhea
* Patients with uncontrolled medical condition(s)
* Patients with a history of non-compliance to oral or injectable medication.
* Patients unwilling to have injectable medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Meltzer, M.D., Principal Investigator — Northwestern University
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred sixty-nine patients who met Diagnostic and Statistical Manual (DSM-IV) criteria for schizophrenia or schizoaffective disorder were screened, and 160 patients were enrolled.
Groups:
- Conventional Dose: All of those who are randomized to the conventional Consta dose will receive it in the form of Consta at a starting dose of 50 mg q 2 weeks (given as two injections - active 50 mg plus placebo injection).
  Subjects will be randomized to conventional dose Consta or high dose Consta. All of those who are randomized to the conventional Consta dose will receive it in the form of Consta at a starting dose of 50 mg q 2 weeks.
- High Dose Group: Those who are randomized to high dose Consta will receive Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose after consent.
  Those who are randomized to high-dose Consta will receive a Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose.
Period: Overall Study
Arm/Group | Conventional Dose | High Dose Group
Started | 82 | 78
Completed | 59 | 55
Not Completed | 23 | 23

BASELINE CHARACTERISTICS:
Groups:
- Conventional Dose: All of those who are randomized to the conventional Consta dose will receive it in the form of Consta at a starting dose of 50 mg q 2 weeks (given as two injections - active 50 mg plus placebo injection).
  long-acting injectable risperidone, Conventional Dose Group: The study dose remains 50 mg for the length of the study.
- High Dose Group: Those who are randomized to high dose Consta will receive Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose after consent.
  long-acting injectable risperidone, High Dose Group: Beginning dose 75 mg. Can be increased to 100 mg at Week 6.
- Total: Total of all reporting groups
Arm/Group | Conventional Dose | High Dose Group | Total
Number analyzed (Participants) | 82 | 78 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 78 | 160
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (10.6) | 41 (11.4) | 40.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 60 | 56 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 76 | 72 | 148
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 82 | 78 | 160

OUTCOME MEASURES:

1. Primary Outcome: Total Positive and Negative Syndrome Scale (PANSS) Score Between Baseline and 24 Weeks.
Description: The mean (SEM) of Positive and Negative Syndrome Scale (PANSS) The Positive and Negative Syndrome Scale (PANSS) is a 30-item questionnaire used to assess the severity of symptoms in schizophrenia. It's considered a gold standard for measuring symptom change in antipsychotic trials and other research. The PANSS is divided into three subscales: positive symptoms, negative symptoms, and general psychopathology. Each item is rated on a 7-point scale, ranging from absent to extreme. Therefore, the minimum possible score of 0 and maximum possible score is 210, but those scores may never be seen in a practical setting. If the score reduces over time that indicates improvement of the symptoms.
Time Frame: six months
Population: patients who met DSM-IV criteria for schizophrenia or schizoaffective disorder
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Conventional Dose: All of those who are randomized to the conventional Consta dose will receive a starting dose of 50 mg q 2 weeks (given as two injections - active 50 mg plus placebo injection).As advised by the package insert for Consta, oral risperidone will be given (3-4 mg qd x 3 days followed by 6mg qd up to Week 3 unless symptoms warrant a quicker titration) along with the injections. Oral risperidone will be discontinued after Week 4. At Week 6, psychopathology will be assessed with PANSS. Dose will remain at 50 mg q 2 weeks for those in the conventional Consta dose group.
- High Dose Group: Those who are randomized to high dose Consta will receive Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose after consent. As advised by the package insert for Consta, oral risperidone will be given (3-4 mg qd x 3 days followed by 6mg qd up to Week 4 unless symptoms warrant a quicker titration) along with the injections. Any oral risperidone the patients receive will be discontinued after Week 4. Psychopathology will be assessed with a PANSS at Week 6. If no improvement since baseline, dose will be increased to two 50 mg injections q 2 weeks for the remainder of the study.
Arm/Group | Conventional Dose | High Dose Group
Number analyzed (Participants) | 82 | 78
score on a scale
  Baseline | 89.0 (1.2) | 89.7 (1.3)
  6 Weeks | 80.0 (1.3) | 80.8 (1.3)
  12 Weeks | 74.2 (1.3) | 78.0 (1.4)
  18 Weeks | 72.3 (1.4) | 74.0 (1.4)
  24 Weeks | 70.9 (1.4) | 72.0 (1.4)

2. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Positive Scale
Description: Positive and Negative Syndrome Scale (PANSS) Positive scale:
  Consists of sum of 7 items, so the score can range from 0 - 49. Improvement means lower scores over time
Time Frame: six months
Population: patients who met DSM-IV criteria for schizophrenia or schizoaffective disorder
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Conventional Dose | High Dose Group
Number analyzed (Participants) | 82 | 78
score on a scale
  PANSS Positive Baseline | 24.0 (0.4) | 24.2 (0.5)
  PANSS Positive 6 Weeks | 20.8 (0.5) | 21.4 (0.5)
  PANSS Positive 12 Weeks | 20.0 (0.5) | 20.0 (0.5)
  PANSS Positive 18 Weeks | 18.2 (0.5) | 19.1 (0.5)
  PANSS Positive 24 Weeks | 18.1 (0.5) | 18.1 (0.5)

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Negative Scale
Description: Positive and Negative Syndrome Scale (PANSS) Negative scale:
  Consists of sum of 7 items, so the score can range from 0 - 49. Improvement means lower scores over time
Time Frame: six months
Population: patients who met DSM-IV criteria for schizophrenia or schizoaffective disorder
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Conventional Dose | High Dose Group
Number analyzed (Participants) | 82 | 78
score on a scale
  PANSS Negative Baseline | 21.0 (0.4) | 21.2 (0.4)
  PANSS Negative 6 Weeks | 19.8 (0.4) | 19.5 (0.4)
  PANSS Negative 12 Weeks | 18.4 (0.4) | 19.2 (0.5)
  PANSS Negative 18 Weeks | 17.9 (0.4) | 18.6 (0.4)
  PANSS Negative 24 Weeks | 17.9 (0.4) | 18.5 (0.5)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Groups:
- Conventional Dose: All of those who are randomized to the conventional Consta dose will receive it in the form of Consta at a starting dose of 50 mg q 2 weeks (given as two injections - active 50 mg plus placebo injection).As advised by the package insert for Consta, oral risperidone will be given (3-4 mg qd x 3 days followed by 6mg qd up to Week 3 unless symptoms warrant a quicker titration) along with the injections.
- High Dose Group: Those who are randomized to high dose Consta will receive Consta 50 mg injection plus 25 mg injection (total dose 75 mg) q 2 weeks as the starting dose after consent. As advised by the package insert for Consta, oral risperidone will be given (3-4 mg qd x 3 days followed by 6mg qd up to Week 4 unless symptoms warrant a quicker titration) along with the injections.
Arm/Group | Conventional Dose | High Dose Group
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/78
Serious Adverse Events (participants affected / at risk) | 2/82 | 5/78
Other Adverse Events (participants affected / at risk) | 14/82 | 13/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Dose (N=82) | High Dose Group (N=78)
Extrapyramidal (Nervous system disorders) | 2 (2) | 5 (5) — Minimal extrapyramidal side effects
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Dose (N=82) | High Dose Group (N=78)
Non-Serious Adverse Events (General disorders) | 14 (19) | 13 (19) — total

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No